CLINICAL TRIAL: NCT02084381
Title: Permeability Enhancement to Reduce Chronic Inflammation _ Medium Cut Off (MCO) (Study no 1502)
Brief Title: PERCI- Medium Cut Off (MCO)
Acronym: PERCI-MCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: German Federal Ministry of Education and Research (Other Government); Gambro Dialysatoren GmbH (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1502
Record Dates: First submitted 2014-02-07; First posted 2014-03-12 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Failure; Chronic Inflammation
Keywords: CKD5, dialysis, high porous membranes
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MCO-Ci 400 (Experimental): MCO-Ci 400 is the investigational medical product applied in hemodialysis mode
  Interventions: Device: MCO-Ci 400
- Revaclear 400 (Active Comparator): the standard high flux dialyzer Revaclear 400 is used as an comparator in hemodialysis mode
  Interventions: Device: Revaclear 400

INTERVENTIONS:
Device: MCO-Ci 400 — hemodialysis
  Arms: MCO-Ci 400
Device: Revaclear 400 — hemodialysis
  Other Names: standard high flux dialyzer
  Arms: Revaclear 400

SUMMARY:
The medium cut-off dialysis membrane has been developed to provide a significantly extended molecular cut-off compared to conventional high-flux membranes. The medium cut-off membrane allows for a high permeability of molecules up to a molecular weight of 45 kDa and has a still limited permeability for albumin (68 kDa).

The main goal of this project is the evaluation of the new, highly porous and selective dialysis membrane (MCO-Ci 400) for the treatment of patients with end-stage renal disease in hemodialysis mode and to study its potential to improve chronic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* CKD5 ( GFR < 15ml/min/ 1.73m2)
* Dialysis treatment for ≥ 3 months
* Dialysis 3x weekly
* Vascular access by fistula or CVC
* Age > 18 and < 99 Years
* Ability to give written informed consent

Exclusion Criteria:

* Missing informed consent form
* current clinically manifested infection or within the last two weeks
* current CRP-value > 50mg/L or within the last two weeks
* Intake of any medication applied for immunosuppressive purposes
* Pregnancy or lactation
* Participation in a different interventional study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
TNF-alpha mRNA | 4 weeks treatment time
  Significant lower pre- dialytic TNF-α mRNA expression level in circulating peripheral blood mononuclear cells

SECONDARY OUTCOMES:
safety related events | 6 month

OTHER OUTCOMES:
Exploratory | 12 weeks
  Elimination of inflammatory molecules and uremic toxins from patient's blood

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Girndt, Prof. Dr., Principal Investigator — Martin-Luther-Universität Halle-Wittenberg
Locations (2):
- Germany (2):
  - Martin-Luther-Universität Halle-Wittenberg, Halle, Saxony-Anhalt
  - Charité - Universitätsmedizin Berlin, Berlin

REFERENCES:
- [Result] Zickler D, Schindler R, Willy K, Martus P, Pawlak M, Storr M, Hulko M, Boehler T, Glomb MA, Liehr K, Henning C, Templin M, Trojanowicz B, Ulrich C, Werner K, Fiedler R, Girndt M. Medium Cut-Off (MCO) Membranes Reduce Inflammation in Chronic Dialysis Patients-A Randomized Controlled Clinical Trial. PLoS One. 2017 Jan 13;12(1):e0169024. doi: 10.1371/journal.pone.0169024. eCollection 2017. PMID 28085888
- [Result] Willy K, Girndt M, Voelkl J, Fiedler R, Martus P, Storr M, Schindler R, Zickler D. Expanded Haemodialysis Therapy of Chronic Haemodialysis Patients Prevents Calcification and Apoptosis of Vascular Smooth Muscle Cells in vitro. Blood Purif. 2018;45(1-3):131-138. doi: 10.1159/000484925. Epub 2017 Dec 22. PMID 29402827
- [Result] Catar R, Moll G, Kamhieh-Milz J, Luecht C, Chen L, Zhao H, Ernst L, Willy K, Girndt M, Fiedler R, Witowski J, Morawietz H, Ringden O, Dragun D, Eckardt KU, Schindler R, Zickler D. Expanded Hemodialysis Therapy Ameliorates Uremia-Induced Systemic Microinflammation and Endothelial Dysfunction by Modulating VEGF, TNF-alpha and AP-1 Signaling. Front Immunol. 2021 Nov 11;12:774052. doi: 10.3389/fimmu.2021.774052. eCollection 2021. PMID 34858433